CLINICAL TRIAL: NCT04442204
Title: Predictors and Mechanisms of Depression and Anxiety During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Omid V. Ebrahimi, Mr., University of Oslo
Other Study IDs: REK125510-10
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective study across two time-points examining the impact of viral mitigation protocols on mental health — Prospective study across two time-points examining the impact of viral mitigation protocols on mental health

SUMMARY:
Study description:

The present study seeks to investigate the predictors and maintaining mechanisms of depression and anxiety symptoms during the COVID-19 pandemic, exactly 3 months following the strictest viral mitigation strategies initiated in Norway in response to the pandemic. This is the time period where the major pandemic protocols are lifted in Norway, following three months of strict pandemic mitigation protocols. The study further aims to identify subgroups with highest levels of depressive and anxiety symptoms during the measurement period, to identify vulnerable subgroups with maintained symptoms three months following the pandemic.

Hypotheses and research questions:

Research Question 1: What is the level of depressive and anxiety symptoms three months following the employment of the strict viral mitigation protocols (i.e., physical distancing protocols) in the general adult population? What are the proportion above the validated cut-offs for depression and general anxiety? Hypothesis 1: There will be a significant decrease in the levels of depression and anxiety symptoms from the baseline (T1) with the strictest mitigation protocols to measurement the measurement period three months into pandemic (T2) where major pandemic mitigation protocols are lifted. Additionally, there will be a significant decrease in the proportion of the sample meeting validated cut-offs for depression and anxiety from T1 to T2.

Hypothesis 2: Higher level at T1 and less reduction from T1 to T2 in positive metacognitions, negative metacognitions, and unhelpful coping strategies all measured with CAS-1, will be related to less reduction in depression and anxiety, above and beyond age, gender, and education. Higher level at T1 and increases from T1 to T2 in physical activity and perceived competence will be related to greater reduction in depression and anxiety, above and beyond, age, gender, and education.

Exploratory: The investigators will further explore the proportion showing reliable change in depression and anxiety and investigate the differences in changes in depression and anxiety across different demographic subgroups in the sample

DETAILED DESCRIPTION:
Hypotheses and research questions:

Research Question 1: What is the level of depressive and anxiety symptoms three months following the employment of the strict viral mitigation protocols (i.e., physical distancing protocols) in the general adult population? What are the proportion above the validated cut-offs for depression and general anxiety? Hypothesis 1: There will be a significant decrease in the levels of depression and anxiety symptoms from the baseline (T1) with the strictest mitigation protocols to measurement the measurement period three months into pandemic (T2) where major pandemic mitigation protocols are lifted. Additionally, there will be a significant decrease in the proportion of the sample meeting validated cut-offs for depression and anxiety from T1 to T2.

Hypothesis 2: Higher level at T1 and less reduction from T1 to T2 in positive metacognitions, negative metacognitions, and unhelpful coping strategies all measured with CAS-1, will be related to less reduction in depression and anxiety, above and beyond age, gender, and education. Higher level at T1 and increases from T1 to T2 in physical activity and perceived competence will be related to greater reduction in depression and anxiety, above and beyond, age, gender, and education.

Explorative: The investigators will further explore the proportion showing reliable change in depression and anxiety and investigate the differences in changes in depression and anxiety across different demographic subgroups in the sample.

Statistical analyses:

Repeated surveys like the present one typically have missing data. Therefore, The investigators will use mixed models instead of paired t-tests, repeated measures ANOVAs, and ordinary linear regression to analyze the data. Mixed models use maximum likelihood estimation, the state of the art approach in handling missing data (Schafer & Graham, 2002). Particularly, if data are missing at random, which is likely in our survey, mixed models present more unbiased results than the other analytic methods (O'Connel et al., 2017). Depression and anxiety will be used as dependent variables in two separate mixed models.

In preliminary analyses, and for each of the dependent variable (PHQ-9; GAD-7), the combination of random effects and covariance structure of residuals that gives the best fit for the "empty" model (the model without fixed predictors except the intercept) will be chosen. Akaike's Information Criterion (AIC) will used to compare the fit of different models. Models that give a reduction in AIC greater than 2 will be considered better (Burnham & Anderson, 2004).

First, H1 about decrease in GAD-7 and PHQ-9 will be investigated by using PHQ-9 (in one analysis) and GAD-7 (in the other) as dependent variable in a model using time (T1 = 0; T2= 1) as a predictor. Second, demographic control variables will be added as predictors. Third, the initial (T1) levels of negative metacognitions, positive metacognitions, unhelpful coping strategies, physical activity, and perceived competence to deal with the crisis, will be added as constant covariates, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the covariates predicting change in anxiety and depression, respectively. Finally, the present (T2) levels of negative metacognitions, positive metacognitions, unhelpful coping strategies, physical activity, and perceived competence to deal with the crisis will be added as constant covariates, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the change in the covariates from T1 to T2 predicting change in depression and anxiety from T1 to T2, respectively.

Descriptive statistics with frequency tables including N, means and SDs and other standard descriptive statistics will examine the research question concerning general levels of depressive- and anxiety symptoms. Subgroup differences will be examined with chi-squared statistics. To investigate the percentage of individuals with depressive and anxiety symptoms, common cut-offs are used; including => 10 on PHQ-9 (Kroenke et al., 2001) and >= 8 on GAD-7 (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).

All analyses and questions addressed in the forthcoming paper that are not pre-specified in this pre-registered protocol will be defined as exploratory.

Sensitivity analyses and random subsample replications of the main findings will be conducted following selection of a random sample of participants that ensure a proportionate ratio between the collected sample and the adult population of Norway.

Possible transformations:

All variables will be assessed in their original and validated format as is recommended practice, as long as this is possible with regards to statistical assumptions underlying the pre-defined analyses (i.e., multiple regression). However, if this is not possible with regards to the statistical assumptions behind the analyses, transformation (e.g., square root or log-transformations) may be needed to apply interval-based methods. The investigators will examine the degree of skewness and evaluate this against the assumptions and analyses before choosing the appropriate analysis. The pre-registered and planned analyses include multiple regression as long as assumptions are met. Alternatively a non-parametric test will be used.

Inference criteria Given the large sample size in this study, the investigators pre-define their significance level: p < 0.01 to determine significance.

Sample size:

The sample size at T1 included a representative and random selection 10 084 adult participants. For the present study at T2, all participants will be invited to participate in accordance with the study plan. The data collection period will continue for up to three weeks until as many of the participants at baseline have responded.

Eligibility criteria:

Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who provide digital consent to partake in the study.

Exclusion Criteria:

* Children and adolescents (individuals below 18)
* Adults not residing in Norway during the measurement period

Measures:

Outcome variables include the following validated measures: PHQ-9 and GAD-7. Predictor variables include the following validated measures: positive metacognitions (measured with CAS-1 subscale); negative metacognitions (measured with CAS-1 subscale); unhelpful coping strategies (also called "strategies"; measured with CAS-1 subscale); physical activity (measure of number of times participant has been physically active for at least 30 minutes in an activity increasing pulse and leading to sweat for the past two weeks); perceived competence to deal with the pandemic (measured with Basic Psychological Needs and Frustration Scale, a single item adapted for the ability to deal pandemic consequences rather than ability to deal with difficult situations in general).

Age, gender and education will be controlled for.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical viral mitigation protocols, and
* Who provide digital consent to partake in the study.

Exclusion Criteria:

* Children and adolescents (individuals below 18)
* Adults not residing in Norway during the measurement period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults residing in Norway experiencing identical mitigation protocols, having equal opportunity of partaking in the survey.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 | Data is set to be collected starting from 22nd of June until enough data has been collected.The data collection period will last no longer than three weeks.
  • The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity, and scores above 10 are considered as the cut-off that indicating that the patient is within the depressive area.
Generalized Anxiety Disorder 7 | Data is set to be collected starting from 22nd of June until enough data has been collected.The data collection period will last no longer than three weeks.
  • The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Specific cut-off for Norwegian samples have been found yielding a cut-off of 8 and above for high sensitivity and specificity (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Omid Ebrahimi, Double PhD Candidate, Principal Investigator — University of Oslo; Asle Hoffart, PhD, Principal Investigator — Modum Bad; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo

REFERENCES:
- [Background] Johnson SU, Ulvenes PG, Oktedalen T, Hoffart A. Psychometric Properties of the General Anxiety Disorder 7-Item (GAD-7) Scale in a Heterogeneous Psychiatric Sample. Front Psychol. 2019 Aug 6;10:1713. doi: 10.3389/fpsyg.2019.01713. eCollection 2019. PMID 31447721
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171